CLINICAL TRIAL: NCT07047209
Title: A Phase 2a Biomarker-Driven Trial of Oral Digoxin in Individuals With Amyotrophic Lateral Sclerosis (ALS) - The Acacia Trial, an ALS MyMatch Trial
Brief Title: Trial of Oral Digoxin in Individuals With Amyotrophic Lateral Sclerosis (ALS)
Acronym: ACACIA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Suma Babu, Study Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P001103
Record Dates: First submitted 2025-06-18; First posted 2025-07-02 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
Keywords: ALS; Amyotrophic Lateral Sclerosis; Early ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Digoxin — Digoxin tablets will be administered orally in a once daily dosage. Each tablet is scored and is of 125 mcg strength. Participants will take 1 tablet, two tablets or half a tablet depending on the dosing tier they are in during study participation.

SUMMARY:
This clinical trial is being conducted to learn about safety and tolerability of digoxin in ALS individuals. Additionally, this trial aims to better understand if digoxin has an effect on slowing neurodegeneration in ALS.

DETAILED DESCRIPTION:
This is a single-arm, Phase 2a, open label, 24-week treatment trial evaluating standard clinical dosages of commercially available, FDA approved oral digoxin in up to 40 eligible ALS participants with early disease (<24 months from symptom onset). The trial will include two cohorts of eligible participants; Cohort 1 of approximately 30 sporadic/non-C9 ALS and Cohort 2 of approximately 10 C9orf72(+) ALS individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent.
2. Adults >18 years of age with a diagnosis of symptomatic ALS as determined by an ALS neurologist, and meets either the revised El Escorial Criteria (clinically possible, probable, probable lab-supported, or definite) or the Gold Coast Criteria.
3. Available or pending CLIA certified ALS genetic panel report.
4. Less than or equal to 24-months since onset of weakness attributed to ALS.
5. Vital capacity (VC) of > 65% predicted value for gender, height and age at screening.
6. Clinically unremarkable Complete Blood Counts, including but not limited to Hemoglobin ≥ 9 g/dL, Platelets ≥ 150 x 109 cells/L.
7. No clinically significant abnormalities in the Comprehensive Metabolic Panel per site/sub-investigator's judgment, including but not limited to:

   1. Serum alanine aminotransferase or aspartate aminotransferase < 3× upper limit of normal, or serum total bilirubin <1.5× upper limit of normal
   2. Estimated GFR (eGFR) of > 30 mL/min/1.73m2
   3. Other clinically significant electrolyte and metabolic abnormalities
8. Ability and willingness to complete all study procedures per the Site Investigator's clinical assessment.
9. Negative pregnancy test within 7 days prior to first dose for women of child-bearing potential (WOCB), defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses any time in the preceding 24 consecutive months).
10. Individuals enrolling in the C9orf72 cohort of the trial must have CLIA certified ALS gene panel demonstrating >31 repeats of C9orf72 hexanucleotide repeat expansion, deemed pathologic.

Exclusion Criteria:

* 1. Clinically significant unstable medical or surgical condition that would pose a risk to the participant's trial procedural participation or interfere with data collection, according to the Site Investigator's judgment (e.g., active infection requiring antibiotics).

  2. Presence of cognitive or mental health disorders impairing ability to provide informed consent for the study per Site investigator assessment.

  3. Active cancer or history of cancer, unless it was successfully treated for durable remission or cure more than 3 years ago. (Note that basal cell carcinoma, squamous cell carcinoma in situ, cervical carcinoma in situ, prostatic carcinoma in situ, or other malignancies that have been curatively excised at any time previously and with no evidence of disease recurrence for at least 3 years are not exclusionary.) 4. Prior solid organ transplantation. 5. Concomitant use of investigational treatments for ALS within 5 half-lives or 30 days, whichever longer.

  6. Screening 12-lead ECG showing QT interval corrected for rate (QTcF) > 470 msec for women and > 450 msec for men, absence of second degree or higher AV block or other clinically significant cardiac arrythmias.

  7. If female, breastfeeding, pregnant, or of child-bearing potential and unwilling to use effective contraception for duration of the trial and after discontinuing treatment.

  8. Serious cardiac condition within the last 6 months, such as uncontrolled arrhythmia, myocardial infarction, unstable angina, or heart disease defined by the New York Heart Association (NYHA) Class III or Class IV or hereditary long QT syndrome.

  9. Exclusion criteria for Lumbar Punctures: active bleeding tendencies OR inability to withhold antiplatelets or anticoagulants safely as per institutional guidelines around LPs OR anatomical spine considerations making it unsafe or challenging for serial LPs OR allergy to local anesthesia used for procedure.

  10. Clinically active cardiac disorders including sinus bradycardia (HR <40 bpm) or sinus tachycardia (HR>140 bpm), cardiac arrythmias [first-degree, second-degree (Wenckebach), or third-degree heart block; atrial tachycardia with block; AV dissociation; accelerated junctional (nodal) rhythm; unifocal or multiform ventricular premature contractions (especially bigeminy or trigeminy); ventricular tachycardia; and ventricular arrythmias]; Persistent or chronic atrial fibrillation that is not controlled using standard medications 11. Concomitant treatment with amiodarone at any dose or quinidine at a dose greater than 20 mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | From drug initiation through study completion, an average of 28 weeks
  Safety: Defined as the occurrence of serious and non-serious treatment-emergent adverse events (TEAEs) and clinically significant treatment-emergent abnormalities in clinical and laboratory values including digoxin trough levels, in ALS individuals treated with study treatment.
Incidence of Completing Study Treatment [Tolerability] | From drug initiation through study completion, an average of 28 weeks
  Tolerability: Defined as percentage of ALS participants who complete the 24 weeks of study treatment, without study drug-attributed intolerable AEs that lead to early permanent drug discontinuation.

SECONDARY OUTCOMES:
Biological Efficacy | From enrollment to the end of study treatment at the Week 24 Visit
  Biological Efficacy: Changes from baseline at week 24 in blood neurofilament light (NfL) levels following oral digoxin treatment.
CNS Penetrance | From enrollment to end of study treatment at the Week 24 Visit
  CNS Penetrance: Defined as CSF digoxin level measurement over 24 weeks of treatment.

OTHER OUTCOMES:
ALS Functional Rating Scale Revised (ALSFRS-R) total and sub-domain scores. | From enrollment to the end of study treatment at the Week 24 Visit
  Changes from baseline at Week 12 and Week 24 in ALS Functional Rating Scale Revised (ALSFRS-R) total and sub-domain scores. The 12 domains included in the ALSFRS-R are rated on a 5-point scale, 0 to 4, with a maximum score of 48 indicating the highest level of functioning.
Slow vital capacity (SVC) | From enrollment to the end of study treatment at the Week 24 Visit
  Changes from baseline at Week 12 and Week 24 in SVC.
Quality of Life measure: ALSAQ-40 total score | From enrollment to the end of study treatment at the Week 24 Visit
  Changes from baseline at Week 12 and Week 24 in ALSAQ-40 scores.
Permanent assisted ventilation-free survival | Permanent assisted ventilation is defined as use of non-invasive or invasive ventilation for >22 hours in a 24-hour period, for 7 consecutive days.
  Changes from baseline at Week 12 and Week 24 in Permanent assisted ventilation-free survival.
Threshold Nerve Conduction Studies | From enrollment to the end of study treatment at the Week 24 Visit.
  Participants at the MGH site will participate in threshold tracking nerve excitability. Evaluate changes from baseline at Week 12 and Week 24 in the electrophysiological endpoints.
CSF analyses of Poly(GP) | From enrollment to the end of study treatment at the Week 24 Visit.
  Fold change from baseline at Week 12 and Week 24 in CSF analyses of biomarkers including poly(GP).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Nova Southeastern University, Davie, Florida
  - Northwestern Universsity, Chicago, Illinois
  - MGH, Boston, Massachusetts